CLINICAL TRIAL: NCT01240915
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled, Parallel Group, Multi-center Study To Investigate The Safety And Efficacy Of Multistem (Pf-05285401) In Subjects With Moderate To Severe Ulcerative Colitis
Brief Title: A Study To Investigate The Safety And Possible Clinical Benefit Of Multistem(r) In Patients With Moderate To Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Healios K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B3041001; 2010-022766-27 (EudraCT Number)
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-01

CONDITIONS: Colitis, Ulcerative
Keywords: safety efficacy MultiStem(r) moderate to severe Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): The first 9 subjects will be recruited into Cohort 1 and will receive either placebo (n=3) or MultiStem low dose (n=6) as an intravenous infusion on Day 1. The first five patients enrolled constitute a subgroup of Cohort 1 and these patients will receive multiple doses, once every day for 7 days for 3 doses (Day 1 and Weeks 1 & 2).
  Interventions: Drug: placebo; Drug: MultiStem low dose
- Cohort 2 (Experimental): This group will receive either placebo (n=3) or MultiStem high dose (n=6) as an intravenous infusion on Day 1. The subjects then receive the opposite dose of study medication at Week 8.
  Interventions: Drug: placebo; Drug: MultiStem high dose
- Cohort 3 (Experimental): These subjects (total n=88 evaluable patients) will receive either Placebo or MultiStem (1:1 randomization) as an intravenous infusion on Day 1. In addition all subjects in Cohort 3 will receive a single infusion of either MultiStem or Placebo at Week 8, depending on their randomization schedule. A total of ~22 patients will receive an additional infusion of MultiStem, ~44 patients will receive the alternative blinded therapy to that which they received for Day 1 infusion, and ~22 patients will receive an additional infusion of placebo.
  Interventions: Drug: placebo; Drug: MultiStem high dose

INTERVENTIONS:
Drug: placebo — once every 7 days for 1- 3 doses
  Arms: Cohort 1
Drug: MultiStem low dose — 1-3 doses
  Arms: Cohort 1
Drug: placebo — Single dose at week 8
  Arms: Cohort 1
Drug: MultiStem low dose — Single dose at week 8
  Arms: Cohort 1
Drug: placebo — Single dose Day 1
  Arms: Cohort 2
Drug: MultiStem high dose — Single dose Day 1
  Arms: Cohort 2
Drug: placebo — Single dose at week 8
  Arms: Cohort 2
Drug: MultiStem high dose — Single dose at week 8
  Arms: Cohort 2
Drug: placebo — Single dose Day 1
  Arms: Cohort 3
Drug: MultiStem high dose — Single dose Day 1
  Arms: Cohort 3
Drug: placebo — Single dose at week 8
  Arms: Cohort 3
Drug: MultiStem high dose — Single dose at week 8
  Arms: Cohort 3

SUMMARY:
MultiStem(r) is a new biological product, manufactured from human stem cells obtained from adult bone marrow or other nonembryonic tissue sources. Factors expressed by MultiStem cells are believed to reduce inflammation and regulate immune system function, protect damaged or injured cells and tissue, promote formation of new blood vessels, and augment tissue repair and healing. MultiStem cell treatment resulted in significant efficacy in a mouse model of Graft versus Host Disease with almost complete reversal of gastrointestinal pathology (similar to pathology that would be expected in Ulcerative Colitis). These data, together with safety data generated in 2 other clinical trials, suggest that MultiStem has the potential to be a new treatment option for patients with ulcerative colitis. This is the first study of MultiStem in this patient population and will cautiously explore the safety/toleration and potential benefit of this new treatment in patients with moderate to severe disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a documented diagnosis of ulcerative colitis at least 6 months prior to screening.
* Subjects must have active moderate-to-severe ulcerative colitis based on Mayo score.
* Subjects must have Modified Baron endoscopic score of at least 2 determined within 7 days of first dosing.
* Subjects must have failed or be intolerant (as determined by the investigator) of at least one of the following treatments for UC: Oral corticosteroids, azathioprine or 6-mercaptopurine (6-MP), or anti-tumor necrosis factor (TNF) therapy, eg, infliximab or adalimumab.
* Subjects must be on stable steroid doses.

Exclusion Criteria:

* Subjects who have abnormal organ and marrow function.
* Subjects with a diagnosis of indeterminate colitis, or clinical findings suggestive of Crohn's disease.
* Subjects who meet Truelove-Witts criteria for severe ulcerative colitis.
* Subjects receiving or who are expected to receive Infliximab or other biologic treatment within 8 weeks of the Day 1 study visit.
* Subjects receiving or who are expected to receive Cyclosporine, mycophenolate, or tacrolimus within 4 weeks of the Day 1 study visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (58):
- United States (37):
  - University of California San Francisco, San Francisco, California
  - USCF Endoscopy Unit at Mount Zion, San Francisco, California
  - Clinical Research of the Rockies, Lafayette, Colorado
  - Rocky Mountain Gastroenterology Associates, LLC, Lakewood, Colorado
  - Arapahoe Gastroenterology, PC, Littleton, Colorado
  - Metropolitan Gastroenterology Group, PC, Washington D.C., District of Columbia
  - Gastroenterology Consultants of Clearwater, Clearwater, Florida
  - West Coast Endoscopy Center, Clearwater, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Jacksonville Center for Endoscopy, Jacksonville, Florida
  - Miami Research Associates, South Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - University of Louisville Healthcare Outpatient Center, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Metropolitan Gastroenterology Group, PC - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Endoscopic Microsurgery Associates, PA, Towson, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Utica Surgery Center, Utica, Michigan
  - Surgery Center of Columbia, Columbia, Missouri
  - Center for Digestive and Liver Diseases, Inc., Mexico, Missouri
  - Present, Chapman, Steinlauf and Marion, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Asher Kornbluth, MD PC, New York, New York
  - Charlotte Gastroenterology and Hepatology, PLLC, Charlotte, North Carolina
  - Wake Internal Medicine Consultants, Inc., Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Wake Forest University University Baptist Medical Center - Internal Medicine, Winston-Salem, North Carolina
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Sentara Leigh Hospital, Norfolk, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - McGuire DVAMC, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Belgium (2):
  - Hopital Erasme / Gastroenterology, Brussels
  - Pfizer Clinical Research Unit, Brussels
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - Northern Alberta Clinical Trials and Research Center, Edmonton, Alberta
  - Zeidler Ledcor Centre - University of Alberta, Edmonton, Alberta
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
- Germany (3):
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Universitaetsklinikum Halle, Halle
  - Medizinische Hochschule Hannover, Hanover
- Hungary (4):
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak/I. Belgyogyaszat es Gastroenterologia, Budapest
  - Pandy Kalman Megyei Korhaz, III. sz. Belosztaly-Gasztroenterologia, Gyula
  - Karolina Korhaz Rendelointezet, Belgyogyaszat, Mosonmagyaróvár
  - Tolna Megyei Balassa Janos Korhaz / II. Belgyogyaszat, Szekszárd
- Italy (3):
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Policlinico Universitario Agostino Gemelli, Roma
- Slovakia (2):
  - Gastroenterologicke a hepatologicke oddelenie, V. interna klinika LFUK a UN Bratislava, Ruzinov, Bratislava, Slovakia
  - Gastroenterologicka ambulancia, GEA s.r.o., Trnava
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset Medicinkliniken, Gothenburg
  - Karolinska Universitetssjukhuset, GastroCentrum Medicin, Stockholm
  - Akademiska sjukhuset, Mag tarmmottagningen, Uppsala

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3041001&StudyName=A%20Study%20To%20Investigate%20The%20Safety%20And%20Possible%20Clinical%20Benefit%20Of%20Multistem%28r%29%20In%20Patients%20With%20Moderate%20To%20Severe%20Ulcerative%20Colit

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Placebo, MultiStem 300: Participants received a single dose (Day 1) or 3 doses (Day 1, Week 1, Week 2) of placebo infusion, followed by a single dose of MultiStem 300 Million Cells infusion at Week 8.
- Cohort 2: Placebo, MultiStem 750; Cohort 3: Placebo, MultiStem 750: Participants received a single dose of placebo infusion on Day 1, followed by a single dose of MultiStem 750 Million Cells infusion at Week 8.
- Cohort 1: MultiStem 300, Placebo: Participants received a single dose of MultiStem 300 Million Cells infusion on Day 1, followed by a single dose of placebo infusion at Week 8.
- Cohort 1: MultiStem 300 (x3), Placebo: Participants received up to 3 doses of MultiStem 300 Million Cells infusion (Day 1, Week, Week 2), followed by a single dose of placebo infusion at Week 8.
- Cohort 2: MultiStem 750, Placebo; Cohort 3: MultiStem 750, Placebo: Participants received a single dose of MultiStem 750 Million Cells infusion on Day 1, followed by a single dose of placebo infusion at Week 8.
- Cohort 3: MultiStem 750, MultiStem 750: Participants received a single dose of MultiStem 750 Million Cells infusion on Day 1, followed by a single dose of MultiStem 750 Million Cells infusion at Week 8.
- Cohort 3: Placebo, Placebo: Participants received a single dose of placebo infusion on Day 1, followed by a single dose of placebo infusion at Week 8.
Period: Overall Study
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Started | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
Completed | 0 | 2 | 2 | 1 | 2 | 13 | 17 | 15 | 13
Not Completed | 2 | 1 | 0 | 3 | 4 | 10 | 8 | 4 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 2 | 0 | 4 | 2 | 3 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Insufficient Clinical Response | 0 | 0 | 0 | 0 | 1 | 3 | 6 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who received at least 1 dose of study medication.
Groups:
- Cohort 1: MultiStem 300 or MultiStem 300 (x3), Placebo: Participants received either a single dose of MultiStem 300 Million Cells infusion on Day 1 or 3 doses on Day 1, Week 1, and Week 2; followed by a single dose of placebo infusion at Week 8.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300 or MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo | Total
Number analyzed (Participants) | 2 | 3 | 6 | 6 | 23 | 25 | 19 | 21 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (7.1) | 52.0 (7.0) | 49.3 (14.1) | 40.0 (14.0) | 43.4 (12.8) | 38.8 (13.4) | 39.8 (12.5) | 42.5 (15.7) | 42.2 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 5 | 7 | 12 | 3 | 7 | 36
  Male | 2 | 2 | 5 | 1 | 16 | 13 | 16 | 14 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Endoscopic Score (as Measured by Modified Baron Score) at Week 8
Description: Modified Baron Score is an instrument designed to measure endoscopic activity of ulcerative colitis. It classifies the mucosal inflammation in 4 grades (0=normal, 1=granular mucosa with an abnormal vascular pattern, 2=friable mucosa, 3=microulceration with spontaneous bleeding, 4=gross ulceration with spontaneous bleeding).
Time Frame: Baseline and Week 8
Population: The full analysis set included all available observed data from all randomized participants who completed at least 1 infusion and were either withdrawn as a treatment failure, or had at least 1 valid post-dose measurement on a primary endpoint. Baseline observation carried forward (BOCF) was used for treatment failures.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Pooled MultiStem: All participants who received MultiStem 750 Million Cells infusion on Day 1 in Cohort 3.
- Pooled Placebo: All participants who received placebo infusion on Day 1 in Cohort 3.
Arm/Group | Pooled MultiStem | Pooled Placebo
Number analyzed (Participants) | 48 | 40
scores on a scale
  Baseline | 3.13 (1.104) | 3.10 (1.128)
  Change at Week 8 | 0.10 (1.134) | -0.30 (1.091)
Statistical Analysis 1: Comparison: Pooled MultiStem vs Pooled Placebo; Pooled MultiStem versus Pooled Placebo; Test type: Superiority or Other; p = 0.96, ANCOVA — 1-sided p-value; Mean Difference (Final Values) = 0.40, 80% CI 2-sided [0.12 to 0.69], Standard Error of Mean 0.223

2. Primary Outcome: Change From Baseline in Rectal Bleeding Mayo Subscore at Week 4
Description: Mayo Score is an instrument designed to measure disease activity of ulcerative colitis. Mayo subscores for rectal bleeding range from 0 to 3, with higher scores indicating more severe disease.
Time Frame: Baseline and Week 4
Population: The full analysis set included all available observed data from all randomized participants who completed at least 1 infusion and were either withdrawn as a treatment failure, or had at least 1 valid post-dose measurement on a primary endpoint; n=the number of participants analyzed at that time point in the respective arms.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pooled MultiStem | Pooled Placebo
Number analyzed (Participants) | 48 | 40
scores on a scale
  Baseline | 1.42 (0.942) | 1.23 (0.832)
  Change at Week 4 | -0.44 (0.943) | -0.38 (0.705)
Statistical Analysis 1: Comparison: Pooled MultiStem vs Pooled Placebo; Pooled MultiStem versus Pooled Placebo (Week 4); Test type: Superiority or Other; p = 0.54, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 8; Mean Difference (Final Values) = 0.02, 80% CI 2-sided [-0.19 to 0.22], Standard Error of Mean 0.161

3. Primary Outcome: Change From Baseline in Rectal Bleeding Mayo Subscore at Week 8
Description: as for outcome 2
Time Frame: Baseline and Week 8
Population: The full analysis set included all available observed data from all randomized participants who completed at least 1 infusion and were either withdrawn as a treatment failure, or had at least 1 valid post-dose measurement on a primary endpoint.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pooled MultiStem | Pooled Placebo
Number analyzed (Participants) | 48 | 40
scores on a scale | -0.46 (1.051) | -0.43 (0.874)
Statistical Analysis 1: Comparison: Pooled MultiStem vs Pooled Placebo; Pooled MultiStem versus Pooled Placebo (Week 8); Test type: Superiority or Other; p = 0.67, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 8; Mean Difference (Final Values) = 0.08, 80% CI 2-sided [-0.15 to 0.30], Standard Error of Mean 0.174

4. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to Week 52
Population: The safety analysis population consisted of all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
participants
  AEs | 2 | 3 | 0 | 4 | 5 | 20 | 18 | 16 | 19
  SAEs | 1 | 0 | 0 | 3 | 0 | 7 | 4 | 5 | 4

5. Primary Outcome: Number of Participants With Treatment-Emergent AEs by System Organ Class (SOC)
Time Frame: Baseline up to Week 52
Population: The safety analysis population consisted of all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
participants
  BLOOD AND LYMPHATIC SYSTEM DISORDERS | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 3 | 4
  CARDIAC DISORDERS | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  EAR AND LABYRINTH DISORDERS | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  ENDOCRINE DISORDERS | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  EYE DISORDERS | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
  GASTROINTESTINAL DISORDERS | 2 | 1 | 0 | 2 | 4 | 13 | 10 | 11 | 12
  GENERAL DISORDERS | 2 | 1 | 0 | 3 | 1 | 8 | 5 | 5 | 6
  IMMUNE SYSTEM DISORDERS | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
  INFECTIONS AND INFESTATIONS | 1 | 1 | 0 | 1 | 1 | 10 | 9 | 9 | 7
  INJURY, POISONING AND PROCEDURAL COMPLICATIONS | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1
  INVESTIGATIONS | 0 | 1 | 0 | 0 | 1 | 4 | 1 | 5 | 3
  METABOLISM AND NUTRITION DISORDERS | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1
  MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS | 0 | 2 | 0 | 0 | 2 | 6 | 5 | 2 | 1
  NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  NERVOUS SYSTEM DISORDERS | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 9 | 6
  PSYCHIATRIC DISORDERS | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2
  RENAL AND URINARY DISORDERS | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS | 1 | 1 | 0 | 0 | 0 | 5 | 5 | 1 | 4
  SKIN AND SUBCUTANEOUS TISSUE DISORDERS | 0 | 0 | 0 | 1 | 1 | 4 | 4 | 3 | 2
  SURGICAL AND MEDICAL PROCEDURES | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  VASCULAR DISORDERS | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 1

6. Primary Outcome: Number of Treatment-Emergent AEs by Severity
Description: The intensity grades were defined as follows: mild=does not interfere with participant's usual function; moderate=interferes to some extent with participant's usual function; severe=interferes significantly with participant's usual function.
Time Frame: Baseline up to Week 52
Population: The safety analysis population consisted of all participants who received at least 1 dose of study medication.
Measure: Number; unit: adverse events
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
adverse events
  Mild AEs | 6 | 16 | 0 | 8 | 13 | 61 | 35 | 56 | 48
  Moderate AEs | 4 | 0 | 0 | 5 | 2 | 33 | 31 | 21 | 17
  Severe AEs | 1 | 0 | 0 | 4 | 0 | 13 | 8 | 4 | 3

7. Secondary Outcome: Change From Baseline in Rectal Bleeding Mayo Subscore at Week 12 and Week 16
Description: as for outcome 2
Time Frame: Baseline, Week 12, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
scores on a scale
  Change at Week 12 (n=0,0,0,0,0,22,25,17,19) | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | -0.77 (0.869) | -0.64 (1.114) | -0.53 (0.874) | -0.47 (0.905)
  Change at Week 16 (n=2,3,2,4,6,21,24,17,19) | -1.50 (0.707) | -1.00 (1.000) | 0.00 (0.000) | 0.00 (0.816) | -0.60 (1.140) | -0.57 (0.978) | -0.92 (1.100) | -0.47 (0.874) | -0.58 (0.838)

8. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: The total number of participants with laboratory test abnormalities with or without regard to baseline abnormality was assessed. Laboratory parameters included: hematology (hemoglobin, hematocrit, red blood cell [RBC] count, platelet count, white blood cell [WBC] count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes, erythrocyte sedimentation rate); chemistry (blood urea nitrogen and creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein; urinalysis (pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, microscopy (only if urine dipstick was positive for blood, protein, nitrites or leukocyte esterase); other (follicle-stimulating hormone, human chorionic gonadotropin, stool microbiology, creatinine kinase, direct bilirubin, indirect bilirubin, gamma-glutamyl transferase, international normalized ratio.
Time Frame: Baseline up to Week 24
Population: The safety analysis population consisted of all participants who received at least 1 dose of study medication; n=the number of participants analyzed at that time point in the respective arms.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
participants
  Normal/Abnormal Baseline(n=2,3,2,4,6,23,25,19,21) | 2 | 2 | 1 | 4 | 4 | 14 | 20 | 15 | 17
  Normal Baseline (n=2,3,2,4,6,23,25,19,21) | 2 | 2 | 1 | 3 | 4 | 9 | 16 | 12 | 13
  Abnormal Baseline (n=2,3,2,2,3,22,19,15,18) | 1 | 1 | 1 | 1 | 2 | 7 | 4 | 4 | 6

9. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Findings
Description: Vital signs assessment included pulse rate, systolic blood pressure (SBP) and diastolic blood pressure (DBP). Criteria for vital sign values meeting potential clinical concern included: SBP <90 millimeters of mercury (mm Hg) and >=30 mm Hg increase/decrease from baseline, DBP <50 mm Hg and >=20 mm Hg increase/decrease from baseline, pulse rate <40 or >120 beats per minute (bpm),
Time Frame: Baseline up to Week 52
Population: The safety analysis population consisted of all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
participants
  Supine SBP <90 mm Hg | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Supine DBP <50 mm Hg | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Supine Pulse Rate <40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine Pulse Rate >120 bpm | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
  Supine SBP >=30 mm Hg Increase From Baseline | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 2
  Supine DBP >=20 mm Hg Increase From Baseline | 2 | 0 | 0 | 1 | 0 | 3 | 0 | 2 | 4
  Supine SBP >=30 mm Hg Decrease From Baseline | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1
  Supine DBP >=20 mm Hg Decrease From Baseline | 1 | 1 | 0 | 0 | 0 | 6 | 1 | 3 | 0

10. Secondary Outcome: Fold Change From Baseline in Fecal Calprotectin at Weeks 4, 8, 12, and 16
Description: Fecal calprotectin, a very stable marker, is a 36kDa calcium and zinc binding protein which is neutrophil-derived. It represents 60% of cytosolic proteins in granulocytes and is a measurement of neutrophil migration to the gastrointestinal tract.
Time Frame: Baseline, Weeks 4, 8, 12 and 16
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: fold change
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
fold change
  Baseline (n=2,3,1,4,5,21,23,19,20) | 690.7549 (17) | 1189.8169 (22) | 739.2300 (NA) — Only 1 participant was analyzed. | 898.2758 (89) | 874.1363 (1462) | 576.5796 (237) | 476.1504 (222) | 513.2139 (208) | 821.1953 (220)
  Change at Week 4 (n=2,3,1,3,5,20,21,18,19) | 0.6297 (50) | 1.8680 (103) | 2.0264 (NA) — Only 1 participant was analyzed. | 2.0549 (112) | 1.0940 (91) | 1.2196 (158) | 0.8179 (314) | 1.0541 (166) | 0.6722 (193)
  Change at Week 8 (n=1,2,1,3,2,18,20,17,20) | 2.4504 (NA) — Only 1 participant was analyzed. | 2.4559 (51) | 2.6199 (NA) — Only 1 participant was analyzed. | 0.5744 (52) | 0.3282 (2) | 1.0704 (220) | 0.7462 (235) | 0.8598 (227) | 0.3479 (242)
  Change at Week 12 (n=0,0,0,0,0,20,21,17,18) | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | 0.9947 (171) | 0.8269 (310) | 0.8788 (293) | 0.5279 (171)
  Change at Week 16 (n=2,3,1,4,4,18,18,16,17) | 2.1672 (49) | 0.7679 (32) | 1.1956 (NA) — Only 1 participant was analyzed. | 0.4459 (139) | 0.2474 (4517) | 0.6473 (277) | 0.8486 (149) | 0.5473 (309) | 0.5275 (243)
Statistical Analysis 1: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo (Week 4); Test type: Superiority or Other; p = 0.53, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 1.02, 80% CI 2-sided [0.73 to 1.42]
Statistical Analysis 2: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo (Week 8); Test type: Superiority or Other; p = 0.91, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 1.48, 80% CI 2-sided [1.02 to 2.14]
Statistical Analysis 3: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 MM versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.81, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 1.38, 80% CI 2-sided [0.86 to 2.23]
Statistical Analysis 4: Comparison: Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, Placebo; Cohort 3 MP versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.44, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 0.94, 80% CI 2-sided [0.59 to 1.51]
Statistical Analysis 5: Comparison: Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 PM versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.67, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 1.18, 80% CI 2-sided [0.72 to 1.94]
Statistical Analysis 6: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 MM versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.62, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 1.12, 80% CI 2-sided [0.68 to 1.84]
Statistical Analysis 7: Comparison: Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, Placebo; Cohort 3 MP versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.95, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 0.95, 80% CI 2-sided [0.58 to 1.57]
Statistical Analysis 8: Comparison: Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 PM versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.30, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 0.81, 80% CI 2-sided [0.49 to 1.36]

11. Secondary Outcome: Fold Change From Baseline in C-Reactive Protein (CRP) at Weeks 4, 8, 12, and 16
Description: CRP is an acute-phase protein which provides an objective criterion of inflammatory activity. CRP has a short half-life (19 hours) and therefore rises early after the onset of inflammation and rapidly decreases after resolution of the inflammation. It is induced by interleukin-6, TNF-alpha and other pro-inflammatory cytokines that are produced within the intestinal lamina propria.
Time Frame: Baseline, Weeks 4, 8, 12 and 16
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: fold change
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
fold change
  Baseline (n=2,3,2,4,6,22,25,19,20) | 1.272 (45) | 1.527 (118) | 0.229 (34) | 0.578 (37) | 0.180 (74) | 0.613 (339) | 0.542 (236) | 0.397 (157) | 0.453 (297)
  Change at Week 4 (n=2,3,2,3,6,21,25,18,20) | 0.289 (9) | 0.555 (82) | 1.937 (42) | 1.285 (60) | 1.446 (54) | 0.891 (147) | 0.764 (140) | 0.999 (103) | 0.588 (132)
  Change at Week 8 (n=1,3,1,3,5,21,25,19,20) | 1.390 (NA) — Only 1 participant was analyzed. | 0.745 (49) | 2.331 (NA) — Only 1 participant was analyzed. | 1.172 (20) | 1.555 (31) | 1.189 (146) | 0.759 (207) | 1.200 (113) | 0.623 (150)
  Change at Week 12 (n=0,0,0,0,0,21,24,17,18) | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | 0.937 (211) | 0.710 (365) | 0.782 (149) | 0.373 (155)
  Change at Week 16 (n=2,3,2,4,5,20,24,17,18) | 0.956 (164) | 0.481 (56) | 0.606 (248) | 0.869 (14) | 1.184 (54) | 0.776 (156) | 0.425 (176) | 0.612 (133) | 0.417 (197)
Statistical Analysis 1: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo (Week 4); Test type: Superiority or Other; p = 0.79, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 1.17, 80% CI 2-sided [0.91 to 1.51]
Statistical Analysis 2: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo (Week 8); Test type: Superiority or Other; p = 0.80, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 1.21, 80% CI 2-sided [0.90 to 1.63]
Statistical Analysis 3: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 MM versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.99, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 2.75, 80% CI 2-sided [1.63 to 4.64]
Statistical Analysis 4: Comparison: Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, Placebo; Cohort 3 MP versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.96, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 1.96, 80% CI 2-sided [1.19 to 3.25]
Statistical Analysis 5: Comparison: Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 PM versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.95, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 1.98, 80% CI 2-sided [1.15 to 3.41]
Statistical Analysis 6: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 MM versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.99, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 2.30, 80% CI 2-sided [1.52 to 3.48]
Statistical Analysis 7: Comparison: Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, Placebo; Cohort 3 MP versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.62, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 1.10, 80% CI 2-sided [0.74 to 1.63]
Statistical Analysis 8: Comparison: Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 PM versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.89, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Geometric Mean Ratio = 1.51, 80% CI 2-sided [0.98 to 2.32]

12. Secondary Outcome: Percentage of Participants With Rectal Bleeding Mayo Subscore of Zero at Weeks 4, 8, 12, and 16
Description: Mayo subscores for rectal bleeding range from 0 to 3 (0=no blood seen; 1=streaks of blood with stool less than half the time; 2=obvious blood with stool most of the time; 3=blood alone passes).
Time Frame: Week 4, 8, 12 and 16
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
percentage of participants
  Week 4 | 50.0 | 66.7 | 50.0 | 33.3 | 40.0 | 52.2 | 28.0 | 31.6 | 42.9
  Week 8 | 50.0 | 66.7 | 50.0 | 33.3 | 40.0 | 47.8 | 36.0 | 31.6 | 47.6
  Week 12 | NA — No participants were analyzed in this arm at Week 12. | NA — No participants were analyzed in this arm at Week 12. | NA — No participants were analyzed in this arm at Week 12. | NA — No participants were analyzed in this arm at Week 12. | NA — No participants were analyzed in this arm at Week 12. | 60.9 | 40.0 | 47.4 | 42.9
  Week 16 | 50.0 | 100 | 50.0 | 50.0 | 40.0 | 47.8 | 48.0 | 36.8 | 52.4
Statistical Analysis 1: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo (Week 4); Test type: Superiority or Other; p = 0.34, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 1.21, 80% CI 2-sided [0.66 to 2.19]
Statistical Analysis 2: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo (Week 8); Test type: Superiority or Other; p = 0.33, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 1.23, 80% CI 2-sided [0.68 to 2.23]
Statistical Analysis 3: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 MM versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.10, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 2.37, 80% CI 2-sided [0.99 to 5.67]
Statistical Analysis 4: Comparison: Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, Placebo; Cohort 3 MP versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.74, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 0.66, 80% CI 2-sided [0.28 to 1.55]
Statistical Analysis 5: Comparison: Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 PM versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.48, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 1.04, 80% CI 2-sided [0.41 to 2.64]
Statistical Analysis 6: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 MM versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.58, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 0.88, 80% CI 2-sided [0.38 to 2.03]
Statistical Analysis 7: Comparison: Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, Placebo; Cohort 3 MP versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.68, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 0.74, 80% CI 2-sided [0.33 to 1.66]
Statistical Analysis 8: Comparison: Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 PM versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.84, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 0.51, 80% CI 2-sided [0.21 to 1.23]

13. Secondary Outcome: Percentage of Participants in Endoscopic Remission at Week 8
Description: Modified Baron Score is an instrument designed to measure endoscopic activity of ulcerative colitis. It classifies the mucosal inflammation in 4 grades (0=normal, 1=granular mucosa with an abnormal vascular pattern, 2=friable mucosa, 3=microulceration with spontaneous bleeding, 4=gross ulceration with spontaneous bleeding). Endoscopic remission is defined as modified Baron Endoscopic Score equal to 0.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
percentage of participants | 0 | 0 | 0 | 0 | 16.7 | 4.3 | 4.0 | 0 | 9.5
Statistical Analysis 1: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo; Test type: Superiority or Other; p = 0.57, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 0.83, 80% CI 2-sided [0.22 to 3.07]

14. Secondary Outcome: Percentage of Participants in Clinical Remission at Week 8
Description: Clinical remission is defined as a total Mayo score of 2 points or lower, with no individual subscores exceeding 1 point.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 8.0 | 0 | 19.0
Statistical Analysis 1: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo; Test type: Superiority or Other; p = 0.85, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 0.39, 80% CI 2-sided [0.12 to 1.23]

15. Secondary Outcome: Percentage of Participants With Decrease From Baseline of at Least 1 Point in Rectal Bleeding Mayo Subscore at Weeks 4, 8, 12, and 16
Description: Mayo subscores for rectal bleeding range from 0 to 3 (0=no blood seen; 1=streaks of blood with stool less than half the time; 2=obvious blood with stool most of the time; 3=blood alone passes). A decrease from baseline score indicates improvement.
Time Frame: Baseline, Weeks 4, 8, 12 and 16
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
percentage of participants
  Week 4 | 100 | 66.7 | 0 | 0 | 40.0 | 43.5 | 48.0 | 21.1 | 38.1
  Week 8 | 100 | 33.3 | 0 | 0 | 40.0 | 34.8 | 48.0 | 31.6 | 47.6
  Week 12 | NA — No participants were analyzed in this arm at Week 12. | NA — No participants were analyzed in this arm at Week 12. | NA — No participants were analyzed in this arm at Week 12. | NA — No participants were analyzed in this arm at Week 12. | NA — No participants were analyzed in this arm at Week 12. | 54.5 | 60.0 | 41.2 | 52.6
  Week 16 | 100 | 66.7 | 0 | 25.0 | 60.0 | 47.6 | 58.3 | 35.3 | 47.4
Statistical Analysis 1: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo (Week 4); Test type: Superiority or Other; p = 0.05, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 2.27, 80% CI 2-sided [1.21 to 4.24]
Statistical Analysis 2: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo (Week 8); Test type: Superiority or Other; p = 0.43, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 1.09, 80% CI 2-sided [0.61 to 1.95]
Statistical Analysis 3: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 MM versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.44, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 1.11, 80% CI 2-sided [0.45 to 2.76]
Statistical Analysis 4: Comparison: Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, Placebo; Cohort 3 MP versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.38, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 1.23, 80% CI 2-sided [0.50 to 3.04]
Statistical Analysis 5: Comparison: Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 PM versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.89, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 0.38, 80% CI 2-sided [0.14 to 1.04]
Statistical Analysis 6: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 MM versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.47, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 1.05, 80% CI 2-sided [0.45 to 2.42]
Statistical Analysis 7: Comparison: Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, Placebo; Cohort 3 MP versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.24, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 1.58, 80% CI 2-sided [0.70 to 3.57]
Statistical Analysis 8: Comparison: Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 PM versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.81, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 0.53, 80% CI 2-sided [0.22 to 1.32]

16. Secondary Outcome: Percentage of Participants With Endoscopic Response at Week 8
Description: Endoscopic response is defined as a decrease in modified Baron endoscopic score from baseline of at least 2 points.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
percentage of participants | 0 | 0 | 0 | 0 | 0 | 8.7 | 8.0 | 10.5 | 19.0
Statistical Analysis 1: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo; Test type: Superiority or Other; p = 0.84, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 0.49, 80% CI 2-sided [0.20 to 1.24]

17. Secondary Outcome: Percentage of Participants in Clinical Response at Week 8
Description: Clinical response is defined as a decrease in total Mayo score from baseline of at least 3 points and at least 30 percent (%), with an accompanying decrease in the subscore for rectal bleeding of at least 1 point or an absolute subscore for rectal bleeding of 0 or 1.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
percentage of participants | 50.0 | 33.3 | 0 | 0 | 0 | 4.3 | 24.0 | 15.8 | 42.9
Statistical Analysis 1: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo; Test type: Superiority or Other; p = 0.96, Regression, Logistic — 1-sided p-value; Odds Ratio (OR) = 0.30, 80% CI 2-sided [0.12 to 0.73]

18. Secondary Outcome: Change From Baseline in Total Mayo Scores at Week 8
Description: Mayo Score is an instrument designed to measure disease activity of ulcerative colitis, with total score ranging from 0 to 12. It consists of 4 subscores (stool frequency, rectal bleeding, findings of flexible proctosigmoidoscopy, and physician global assessment [PGA]), each graded from 0 to 3, with higher scores indicating more severe disease.
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
scores on a scale
  Baseline (n=2,3,2,4,6,23,25,19,21) | 10.00 (2.828) | 7.33 (1.155) | 8.50 (0.707) | 7.75 (0.957) | 7.50 (2.258) | 8.74 (1.839) | 8.48 (2.143) | 8.47 (1.806) | 8.14 (2.220)
  Change at Week 8 (n=2,3,2,3,5,23,25,19,21) | -2.00 (1.414) [-1.84 to 0.33] | 0.00 (2.646) [-2.32 to -0.30] | 1.00 (1.414) [-2.11 to 0.18] | 0.33 (0.577) [-3.37 to -1.15] | -0.60 (0.894) | -0.78 (2.088) | -1.20 (2.872) | -0.89 (2.132) | -2.00 (2.683)
Statistical Analysis 1: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo; Test type: Superiority or Other; p = 0.87, ANCOVA — 1-sided p-value; Mean Difference (Final Values) = 0.58, 80% CI 2-sided [-0.08 to 1.24], Standard Error of Mean 0.513

19. Secondary Outcome: Change From Baseline in Partial Mayo Scores at Weeks 4, 8, 12, and 16
Description: Mayo Score is an instrument designed to measure disease activity of ulcerative colitis. Mayo Score ranges from 0 to 12 points. It consists of 4 subscores, each graded from 0 to 3 with higher scores indicating more severe disease. A Partial Mayo Score (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and calculated as the sum of 3 subscores (stool frequency, rectal bleeding and PGA) with each ranging from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). Higher scores indicate more severe disease.
Time Frame: Baseline, Weeks 4, 8, 12 and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
scores on a scale
  Baseline (n=2,3,2,4,6,23,25,19,21) | 7.50 (2.121) | 5.33 (0.577) | 6.00 (1.414) | 5.75 (0.500) | 5.50 (1.378) | 6.22 (1.347) | 6.08 (1.605) | 6.00 (1.202) | 5.71 (1.736)
  Change at Week 4 (n=2,3,2,3,5,23,25,19,21) | -3.00 (0.000) [-1.84 to 0.33] | -2.00 (1.732) [-2.32 to -0.30] | -0.50 (0.707) [-2.11 to 0.18] | 0.67 (1.528) [-3.37 to -1.15] | -0.40 (1.140) | -1.00 (1.414) | -0.96 (1.791) | -1.16 (1.675) | -1.24 (1.895)
  Change at Week 8 (n=2,3,2,3,5,23,25,19,21) | -2.00 (1.414) | -1.00 (1.732) | 0.50 (0.707) | 0.33 (0.577) | -0.80 (1.095) | -0.91 (1.756) | -1.12 (2.472) | -0.79 (1.653) | -1.62 (2.037)
  Change at Week 12 (n=0,0,0,0,0,22,25,17,19) | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | NA (NA) — No participants were analyzed in this arm at Week 12. | -1.91 (1.974) | -1.52 (2.312) | -2.06 (2.135) | -2.11 (2.622)
  Change at Week 16 (2,3,2,4,5,21,24,17,19) | -1.50 (0.707) | -3.00 (3.000) | -1.00 (2.828) | -1.25 (3.403) | -2.20 (1.924) | -1.86 (2.081) | -2.54 (2.621) | -2.41 (2.181) | -2.63 (2.033)
Statistical Analysis 1: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo (Week 4); Test type: Superiority or Other; p = 0.80, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = 0.29, 80% CI 2-sided [-0.15 to 0.74], Standard Error of Mean 0.345
Statistical Analysis 2: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo (Week 8); Test type: Superiority or Other; p = 0.77, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = 0.30, 80% CI 2-sided [-0.23 to 0.84], Standard Error of Mean 0.418
Statistical Analysis 3: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 MM versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.74, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = 0.44, 80% CI 2-sided [-0.42 to 1.30], Standard Error of Mean 0.666
Statistical Analysis 4: Comparison: Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, Placebo; Cohort 3 MP versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.88, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = 0.76, 80% CI 2-sided [-0.08 to 1.59], Standard Error of Mean 0.645
Statistical Analysis 5: Comparison: Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 PM versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.72, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = 0.42, 80% CI 2-sided [-0.50 to 1.33], Standard Error of Mean 0.705
Statistical Analysis 6: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 MM versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.97, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = 1.21, 80% CI 2-sided [0.37 to 2.06], Standard Error of Mean 0.656
Statistical Analysis 7: Comparison: Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, Placebo; Cohort 3 MP versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.75, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = 0.43, 80% CI 2-sided [-0.39 to 1.25], Standard Error of Mean 0.635
Statistical Analysis 8: Comparison: Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 PM versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.85, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = 0.73, 80% CI 2-sided [-0.16 to 1.63], Standard Error of Mean 0.692

20. Secondary Outcome: Change From Baseline in Biopsy Histology Scores at Week 8
Description: A 15 to 25 centimeter (cm) biopsy sample of inflamed mucosal tissue was taken from the worst affected area and scored using the Riley Index. The Riley Index is a histologic scoring system for the assessment of the activity and severity of ulcerative colitis, ranging from 0 to 24. It consists of 6 histologic features (acute inflammatory cell infiltrate, crypt abscesses, mucin depletion, surface epithelial integrity, chronic inflammatory cell infiltrate, and crypt architectural irregularities), all scored on a 4-point scale (higher scores indicate more severe disease).
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
scores on a scale
  Baseline(n=2,3,2,4,5,22,24,18,21) | 9.0 (1.41) | 9.7 (3.79) | 11.0 (2.83) | 7.0 (3.92) | 10.8 (3.77) | 9.4 (4.37) | 10.4 (4.24) | 9.9 (4.17) | 9.7 (5.14)
  Change at Week 4 (n=2,3,1,3,5,21,24,15,20) | -3.5 (4.95) [-1.84 to 0.33] | 1.3 (1.15) [-2.32 to -0.30] | -3.0 (NA) [-2.11 to 0.18] — No standard deviation was calculated, as only 1 participant was analyzed. | -1.0 (1.73) [-3.37 to -1.15] | -0.4 (2.07) | 1.4 (4.63) | -1.0 (3.76) | 0.9 (4.09) | -1.5 (4.80)
Statistical Analysis 1: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo; Test type: Superiority or Other; p = 0.75, ANCOVA — 1-sided p-value; Mean Difference (Final Values) = 0.52, 80% CI 2-sided [-0.46 to 1.49], Standard Error of Mean 0.753

21. Secondary Outcome: Change From Baseline in Patient-Reported Rectal Bleeding up to Week 16
Description: Patient-reported diary data assessed the number of bowel movements (BM) per day when not having a flare and the presence of blood in the stools (rectal bleeding [RB]), if any.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Number analyzed (Participants) | 2 | 3 | 2 | 4 | 6 | 23 | 25 | 19 | 21
scores on a scale
  BM: Baseline(n=2,3,2,4,6,23,25,19,21) | 12.50 (4.950) | 8.00 (2.784) | 6.75 (2.475) | 11.75 (10.508) | 8.42 (3.089) | 7.50 (3.490) | 7.78 (3.781) | 7.50 (3.571) | 6.88 (4.886)
  BM: Change at Week 1 (n=2,3,2,4,5,23,25,19,21) | -1.60 (2.263) [-1.84 to 0.33] | -1.89 (1.766) [-2.32 to -0.30] | 4.15 (2.845) [-2.11 to 0.18] | -0.60 (2.177) [-3.37 to -1.15] | 0.40 (1.300) | -0.42 (1.509) | -0.59 (1.657) | -0.56 (1.215) | -0.81 (3.421)
  BM: Change at Week 4 (n=2,2,2,3,5,23,23,16,19 | -1.43 (3.435) | -1.89 (5.101) | 2.36 (0.505) | 0.17 (2.038) | 1.31 (1.432) | -0.81 (2.088) | 0.28 (3.956) | -0.63 (1.856) | -1.08 (2.575)
  BM: Change at Week 8 (n=2,3,2,3,6,23,23,16,19) | -1.67 (3.771) | -0.86 (3.517) | 3.18 (0.758) | 0.17 (2.754) | 0.41 (2.131) | -0.89 (2.864) | -1.15 (2.833) | 0.18 (2.531) | -1.41 (3.208)
  BM: Change at Week 12 (n=1,1,1,2,2,21,25,16,18) | 0.14 (NA) — No standard deviation was calculated as only 1 participant was analyzed. | 1.43 (NA) — No standard deviation was calculated as only 1 participant was analyzed. | 1.57 (NA) — No standard deviation was calculated as only 1 participant was analyzed. | -1.68 (2.374) | 0.00 (0.000) | -0.67 (3.152) | -0.59 (4.426) | -1.77 (2.301) | -2.02 (3.502)
  BM: Change at Week 16 (n=1,3,2,3,4,22,24,16,18) | 0.00 (NA) — No standard deviation was calculated as only 1 participant was analyzed. | -2.51 (3.716) | 1.72 (0.596) | -0.12 (2.324) | -2.45 (2.208) | -1.81 (3.278) | -2.17 (3.523) | -1.68 (2.899) | -1.86 (3.616)
  RB: Baseline (n=2,3,2,4,6,23,25,19,21) | 1.25 (1.061) | 1.17 (1.258) | 1.00 (1.414) | 1.00 (0.816) | 1.33 (0.816) | 1.20 (0.974) | 1.46 (0.978) | 0.97 (0.950) | 1.05 (0.820)
  RB: Change at Week 1 (n=2,3,2,4,5,23,25,19,21) | -0.32 (0.253) | -1.00 (1.167) | -0.33 (0.471) | -0.12 (0.158) | -0.30 (0.415) | -0.36 (0.697) | -0.24 (0.605) | -0.05 (0.574) | -0.10 (0.408)
  RB: Change at Week 4 (n=2,2,2,3,5,23,23,16,19) | -0.75 (0.354) | -0.29 (1.010) | -0.25 (0.354) | 0.14 (0.378) | -0.71 (0.990) | -0.34 (0.883) | -0.47 (0.840) | -0.27 (0.738) | -0.26 (0.604)
  RB: Change at Week 8 (n=2,3,2,3,6,22,23,13,20) | -0.75 (0.354) | -0.50 (0.500) | 0.00 (0.000) | 0.33 (0.577) | -0.47 (1.035) | -0.40 (0.709) | -0.51 (0.805) | -0.19 (0.997) | -0.51 (0.967)
  RB: Change at Week 12 (n=1,1,1,2,2,21,25,16,18) | -0.57 (NA) — No standard deviation was calculated as only 1 participant was analyzed. | 0.00 (NA) — No standard deviation was calculated as only 1 participant was analyzed. | 0.00 (NA) — No standard deviation was calculated as only 1 participant was analyzed. | 0.00 (0.000) | 0.00 (0.000) | -0.60 (0.792) | -0.49 (1.084) | -0.48 (0.829) | -0.39 (0.783)
  RB: Change at Week 16 (n=1,3,2,3,4,22,24,16,18) | -1.00 (NA) — No standard deviation was calculated as only 1 participant was analyzed. | -1.17 (1.258) | -0.10 (0.141) | 0.33 (0.577) | -1.14 (0.865) | -0.41 (0.936) | -0.86 (1.106) | -0.41 (0.838) | -0.39 (0.874)
Statistical Analysis 1: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo (Week 4); Test type: Superiority or Other; p = 0.51, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = 0.00, 80% CI 2-sided [-0.18 to 0.19], Standard Error of Mean 0.144
Statistical Analysis 2: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Pooled MultiStem versus Pooled Placebo (Week 8); Test type: Superiority or Other; p = 0.62, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = 0.05, 80% CI 2-sided [-0.16 to 0.25], Standard Error of Mean 0.158
Statistical Analysis 3: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 MM versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.29, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = -0.12, 80% CI 2-sided [-0.39 to 0.16], Standard Error of Mean 0.213
Statistical Analysis 4: Comparison: Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, Placebo; Cohort 3 MP versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.74, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = 0.13, 80% CI 2-sided [-0.14 to 0.40], Standard Error of Mean 0.209
Statistical Analysis 5: Comparison: Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 PM versus Cohort 3 PP (Week 12); Test type: Superiority or Other; p = 0.36, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = -0.08, 80% CI 2-sided [-0.37 to 0.21], Standard Error of Mean 0.226
Statistical Analysis 6: Comparison: Cohort 3: MultiStem 750, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 MM versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.56, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = 0.04, 80% CI 2-sided [-0.26 to 0.34], Standard Error of Mean 0.234
Statistical Analysis 7: Comparison: Cohort 3: MultiStem 750, Placebo vs Cohort 3: Placebo, Placebo; Cohort 3 MP versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.18, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = -0.21, 80% CI 2-sided [-0.51 to 0.09], Standard Error of Mean 0.231
Statistical Analysis 8: Comparison: Cohort 3: Placebo, MultiStem 750 vs Cohort 3: Placebo, Placebo; Cohort 3 PM versus Cohort 3 PP (Week 16); Test type: Superiority or Other; p = 0.31, Mixed Models Analysis — 1-sided p-value; MMRM using data up to Week 16; Mean Difference (Final Values) = -0.12, 80% CI 2-sided [-0.45 to 0.20], Standard Error of Mean 0.250

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last study drug administration.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or 1 participant may have experienced both an AE and SAE during the study. All treated participants were included in the analysis.
Arm/Group | Cohort 1: Placebo, MultiStem 300 | Cohort 2: Placebo, MultiStem 750 | Cohort 1: MultiStem 300, Placebo | Cohort 1: MultiStem 300 (x3), Placebo | Cohort 2: MultiStem 750, Placebo | Cohort 3: MultiStem 750, MultiStem 750 | Cohort 3: MultiStem 750, Placebo | Cohort 3: Placebo, MultiStem 750 | Cohort 3: Placebo, Placebo
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/3 | 0/2 | 3/4 | 0/6 | 7/23 | 4/25 | 5/19 | 4/21
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 0/2 | 3/4 | 5/6 | 18/23 | 16/25 | 15/19 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Placebo, MultiStem 300 (N=2) | Cohort 2: Placebo, MultiStem 750 (N=3) | Cohort 1: MultiStem 300, Placebo (N=2) | Cohort 1: MultiStem 300 (x3), Placebo (N=4) | Cohort 2: MultiStem 750, Placebo (N=6) | Cohort 3: MultiStem 750, MultiStem 750 (N=23) | Cohort 3: MultiStem 750, Placebo (N=25) | Cohort 3: Placebo, MultiStem 750 (N=19) | Cohort 3: Placebo, Placebo (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 5 | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Superior sagittal sinus thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diastolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cohort 1: Placebo, MultiStem 300 (N=2) | Cohort 2: Placebo, MultiStem 750 (N=3) | Cohort 1: MultiStem 300, Placebo (N=2) | Cohort 1: MultiStem 300 (x3), Placebo (N=4) | Cohort 2: MultiStem 750, Placebo (N=6) | Cohort 3: MultiStem 750, MultiStem 750 (N=23) | Cohort 3: MultiStem 750, Placebo (N=25) | Cohort 3: Placebo, MultiStem 750 (N=19) | Cohort 3: Placebo, Placebo (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 3 | 5
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 2
Painful defaecation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Perianal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 2
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 3 | 0 | 2 | 2 | 1 | 2
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 5 | 4
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Antibody test (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial test (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cold agglutinins (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0/2 | 0 | 0/0 | 0/1 | 0/16 | 0/13 | 0/16 | 1/14
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 7 | 6
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileostomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.